CLINICAL TRIAL: NCT03656367
Title: Designing Biofunctional Dairy Foods: Matrix Structure of Dairy Products in Relation to Lipaemia
Acronym: DAIRYMAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Birgitte Raben (Other)
Collaborators: University of Aarhus (Other); Arla Foods (Industry)
Responsible Party: Sponsor-Investigator, Anne Birgitte Raben, professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: B346 (H-18024447)
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Lipaemia
Keywords: glycaemia; insulinemia; lipaemia; appetite
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the characteristics of the study design, blinding of project personnel and participants is not possible. However, statistical analyses of the results will be performed in a blinded fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- All subjects (Experimental): Cross-over study (all subjects receive all interventions)
  * Cheddar cheese
  * Blended and homogenized cheddar cheese
  * An analog milk
  * An analog cheese
  Interventions: Dietary Supplement: Cheddar cheese; Dietary Supplement: Blended and homogenized cheddar cheese; Dietary Supplement: An analog milk; Dietary Supplement: An analog cheese
- Healthy subjects only (subgroup) (Other): If any subjects (against our hypothesis) have indices of metabolic syndrome i.e. raised fasting glucose or TG concentration, secondary analyses will be conducted to assess results without these subjects.
  All subjects receive all interventions)
  * Cheddar cheese
  * Blended and homogenized cheddar cheese
  * An analog milk
  * An analog cheese
  Interventions: Dietary Supplement: Cheddar cheese; Dietary Supplement: Blended and homogenized cheddar cheese; Dietary Supplement: An analog milk; Dietary Supplement: An analog cheese

INTERVENTIONS:
Dietary Supplement: Cheddar cheese — The reference product is a commercial matured cheddar cheese
Dietary Supplement: Blended and homogenized cheddar cheese — A blended and homogenized cheddar cheese (a spread) which, compared to the reference, has a minimal protein network and has smaller fat droplet
Dietary Supplement: An analog milk — An anolog milk (i.e. milk with a cheese-like nutritional composition) which, compared to the reference, does not contain a protein network
Dietary Supplement: An analog cheese — This analog cheese (a gel/yoghurt) is produced from the analog milk which, compared to the reference, has a protein network, however it is a network that differs from the reference

SUMMARY:
The overall aim of this study is to investigate how dairy products with different structures and textures affect lipid absorption kinetics in the acute postprandial period via blood lipid biochemistry.

The study will be conducted as a randomized acute cross-over meal study. Apparently healthy men will be recruited in the study. They will on 4 test days consume the 4 dairy products and blood will be drawn the following 8 hours.

DETAILED DESCRIPTION:
The overall aim of this study is to investigate how dairy products with similar nutrient content but different structures and textures affect lipid absorption kinetics in the acute postprandial period via blood lipid biochemistry, as well as nuclear magnetic resonance (NMR) and liquid chromatography mass spectrometry (LCMS)-based metabolomics.

The study will be conducted as a randomized acute cross-over meal study. On four different test days (with a minimum of 2 weeks washout period) four dairy products with similar nutrient composition but different structures or textures will be tested. During each meal test a single dairy product (+ bread and water) is served and postprandial blood samples are collected the following 8 hours. Subjective appetite measurements (VAS) are filled in during the 8-hour period and an ad libitum meal is served in the end of the day.

25 apparently healthy men (weight stable, 18-40 years, 18.5-24.9 kg/m2) will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men
* 18-40 years of age
* Body mass index (BMI): 18.5-24.9 kg/m^2
* Non-smoker
* Haemoglobin concentration ≥8.4 mmol/L

Exclusion Criteria:

* Dislike for dairy products such as milk, cheese and yoghurt
* Weight change >3 kg 2 months prior to study
* Any other blood donation < 3 month prior to study and during study, than the blood donation that is included in this study
* Intensive physical training (>10 hours of per week)
* Self-reported eating disorders or irregular eating schedules (e.g. skipping breakfast) and uncommon diets (vegetarians, vegans etc.)
* Alcohol intake above the recommendation from the Danish Health and Medicines Authority (>21 units of alcohol per week)
* Night- or shift work
* Food intolerance and allergies related to test products e.g. lactose and gluten
* Dietary supplements, if not taken on a regular basis
* Currently use, or use within previously 3 months of prescription medication, except non-prescription primary analgetica (NSAID and paracetamol) to relieve e.g. head ache and stomach pain, and glucocorticoider for topical use e.g. in ointment and creams.
* Chronic diseases e.g. cancer within the past 5 years (except adequately-treated localized basal cell skin cancer), asthma, back pain, thyroid disease, heart disease, diabetes, inflammation
* Disorders: neurological, sleep, diagnosed psychiatric disorder, and gastro intestinal and liver disorders.
* Surgical treatment of obesity and abdominal surgery
* Inability, physically or mental, to comply with the procedures required by the study protocol as evaluated by the daily study manager, principal investigator or clinical responsible
* Subject's general condition contraindicates continuing the study as evaluated by the daily study manager, principal investigator or clinical responsible
* Simultaneous participation in other clinical intervention studies

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Triglyceride | 0-8 hour
  The sample size is calculated on this endpoint. Fasting and postprandial concentrations of triglycerides (mmol/L) are measured after intake of a test meal.
Apolipoprotein B48 | 0-8 hour
  Co-primary endpoint. Fasting and postprandial concentrations of apolipoprotein B48 are measured after intake of a test meal.

SECONDARY OUTCOMES:
Cholesterol (total, LDL and HDL cholesterol) | 0-8 hour
  Fasting and postprandial concentrations of cholesterol (mmol/L) are measured after intake of a test meal.
Free Fatty Acid (FFA) | 0-8 hour
  Fasting and postprandial concentrations of FFA (umol/L) are measured after intake of a test meal.
Insulin | 0-8 hour
  Fasting and postprandial concentrations of insulin (pmol/L) are measured after intake of a test meal.
Glucose | 0-8 hour
  Fasting and postprandial concentrations of glucose (mmol/L) are measured after intake of a test meal.
Apolipoproteins | 0-8 hour
  Fasting and postprandial concentrations of apolipoproteins (e.g. B100) are measured after intake of a test meal.

OTHER OUTCOMES:
Paracetamol | 0-8 hour
  Gastric emptying rate is evaluated by paracetamol (measured as fasting and postprandial concentrations after intake of a test meal).
Metabolomics | 0-8 hour
  Detailed absorption kinetics will be evaluated by NMR-based metabolomics
Subjective appetite sensation | 0-8 hour
  Subjective appetite sensation (e.g. hunger, satiety, thirst) will be evaluated by visual analogue scales (VAS). The VAS is a line (100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating of the subject's sensations. For example, Q: "How hungry do you feel now?", rating: "not at all" (=0 mm) and "extremely" (=100 mm)
Acute energy intake | 8 hours after test meal
  Acute energy intake is evaluated by energy intake of an ad libitum meal that is served after the 8-hour test meal period
Appetite hormones | 0-8 hour
  Fasting and postprandial concentrations of appetite hormones (e.g. GLP-1) may be measured after intake of a test meal.
detailed metabolomics | 0-8 hour
  Detailed absorption kinetics will be evaluated by LCMS-based metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Anne B Raben, prof, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, Frederiksberg, Denmark

REFERENCES:
- [Result] Kjolbaek L, Schmidt JM, Rouy E, Jensen KJ, Astrup A, Bertram HC, Hammershoj M, Raben A. Matrix structure of dairy products results in different postprandial lipid responses: a randomized crossover trial. Am J Clin Nutr. 2021 Nov 8;114(5):1729-1742. doi: 10.1093/ajcn/nqab220. PMID 34477812
- [Result] Thogersen R, Lindahl IEI, Khakimov B, Kjolbaek L, Juhl Jensen K, Astrup A, Hammershoj M, Raben A, Bertram HC. Progression of Postprandial Blood Plasma Phospholipids Following Acute Intake of Different Dairy Matrices: A Randomized Crossover Trial. Metabolites. 2021 Jul 14;11(7):454. doi: 10.3390/metabo11070454. PMID 34357348
- [Result] Schmidt JM, Kjolbaek L, Jensen KJ, Rouy E, Bertram HC, Larsen T, Raben A, Astrup A, Hammershoj M. Influence of type of dairy matrix micro- and macrostructure on in vitro lipid digestion. Food Funct. 2020 Jun 24;11(6):4960-4972. doi: 10.1039/d0fo00785d. PMID 32500911